CLINICAL TRIAL: NCT00576732
Title: Risperidone in the Treatment of Children and Adolescents With Autistic Disorder: A Double-Blind, Placebo-Controlled Study of Efficacy and Safety, Followed by an Open-Label Extension Study of Safety
Brief Title: A Study of the Effectiveness and Safety of Two Doses of Risperidone in the Treatment of Children and Adolescents With Autistic Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CR014740; RISAUT4002
Record Dates: First submitted 2007-12-17; First posted 2007-12-19 (Estimated); Results first posted 2010-09-28 (Estimated); Last update posted 2014-05-09 (Estimated); Status verified 2014-04

CONDITIONS: Autistic Disorder; Autism
Keywords: Irritability; Risperidone; Antipsychotic agent; Autism; Adolescents; Children
MeSH Terms: conditions — Autistic Disorder | interventions — Risperidone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 001 (Experimental): Risperidone low dose Risperidone oral solution 0.125 mg (if <45 kg) or 0.175 mg (if >=45 kg) qd or bid for 6 weeks
  Interventions: Drug: Risperidone low dose
- 002 (Experimental): Risperidone high dose Risperidone oral solution 1.25 mg (if <45 kg) or 1.75 mg (if >=45 kg) qd or bid for 6 weeks
  Interventions: Drug: Risperidone high dose
- 003 (Placebo Comparator): Placebo Oral solution qd or bid for 6 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Oral solution qd or bid for 6 weeks
  Arms: 003
Drug: Risperidone high dose — Risperidone oral solution 1.25 mg (if <45 kg) or 1.75 mg (if >=45 kg) qd or bid for 6 weeks
  Arms: 002
Drug: Risperidone low dose — Risperidone oral solution 0.125 mg (if <45 kg) or 0.175 mg (if >=45 kg) qd or bid for 6 weeks
  Arms: 001

SUMMARY:
The purpose of this study is to evaluate the effectiveness (change in level of irritability and related behaviors) and safety and tolerability of the administration of 2 different fixed dose levels of risperidone (an atypical antipsychotic drug) compared with placebo in children or adolescents who have autism, and to evaluate the safety and tolerability of the drug for additional 26 weeks after the initial 6-week study period.

DETAILED DESCRIPTION:
Autistic Disorder is a condition that develops early in childhood and persists throughout life. Seventy-five percent of children and adolescents with autistic disorder have irritability symptoms such as aggression towards others, deliberate self-injurious behavior, temper tantrums, and quickly changing moods. These symptoms affect their daily functioning such as school performance, interactions with family members and compliance to treatment. Risperidone is an atypical antipsychotic agent that has been recently approved for the treatment of irritability associated with Autistic Disorder in children and adolescents aged 5 to 16 years. The approved dose range is 0.5-3 mg per day. The aim of this study is to evaluate the effectiveness (change in level of irritability and related behaviors) of a lower dose (0.125 mg or 0.175 mg risperidone per day depending on body weight). The study will include three treatment groups. A placebo group, a low dose risperidone group and a higher dose risperidone group (1.25 mg or 1.75mg per day depending on body weight). This phase of the study will be 6 weeks. During the study, neither investigators nor the patients will be told which treatment the patient received. This is called "double blind". The placebo treatment is not expected to be effective. The higher dose group is expected to be effective. At the end of the study, data from the lower dose group will be compared to the placebo group to see if it is effective. Another aim of this study is to evaluate the safety and tolerability of risperidone. At the end of the 6-week double-blind period, patients may enter a 6-month open-label period during which all patients will receive risperidone. During this phase of the study, the doses can be adjusted to a maximum of 1.25 mg or 1.75mg per day depending on body weight. Both investigator and the patient will know what dose the patient is taking. About 93 patients will be randomized. The study will be conducted by investigators from about 15 clinics. Assessments of effectiveness include the Aberrant Behavior Checklist (ABC) subscales including the irritability subscale (ABC-I), the Clinical Global Impression of Change (CGI C); the Clinical Global Impression of Severity (CGI-S); the response rate, and the Compulsions Subscale of the Children's Yale-Brown Obsessive Compulsive Scale (CY BOCS). Safety evaluations include monitoring of adverse events, physical examinations, clinical laboratory tests, nighttime sleep quality and daytime drowsiness, and extrapyramidal symptoms (EPS) as assessed using the Abnormal Involuntary Movement Scale (AIMS), the Barnes Akathisia Rating Scale (BARS) and the Simpson-Angus Scale (SAS). Venous blood samples will be collected for the determination of plasma concentrations of risperidone and 9-hydroxyrisperidone. The study hypotheses are that the higher dose level of risperidone is significantly superior to placebo as measured by change from baseline on the ABC-I Subscale score at end point (Week 6 or early withdrawal) and that the lower dose level of risperidone is significantly superior to placebo as measured by change from baseline on the ABC-I Subscale score at end point (Week 6 or early withdrawal). Double-blind phase: Risperidone oral solutions taken once daily. Depending on body weight patients take 1.25 mL or 1.75 mL of either a 0.1 mg/mL or a 1.0 mg/mL risperidone solution or matching placebo, for 6 weeks. Open-label phase: Medication can be taken once or twice a day. Starting from 0.125mg or 0.175mg per day, drug levels are titrated over 2 weeks to a maximum dose level of 1.25 mg risperidone/day or 1.75 mg /day depending on body weight, for 26 weeks.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV diagnosis of Autistic Disorder (299.00)
* ABC-I Subscale score of greater than or equal to 18
* CGI-S of greater than or equal to 4
* mental age >18 months, body weight of at least 20 kg, seizure-free for at least 6 consecutive months and if on anticonvulsants must be on a dosage that has been stable for at least 4 weeks
* Medication free for 1 week before the start of the study for all psychotropic drugs, except 4 weeks for fluoxetine and at least 8 weeks for injectable medications
* Female patients must be premenarchal or sexually abstinent or, if heterosexually active, must practice an effective method of birth control.

Exclusion Criteria:

* History of prior or current DSM-IV psychotic disorder (e.g., schizophrenia, bipolar disorder, other psychosis), Pervasive Developmental Disorder not otherwise specified (PDD NOS), Asperger's, or Rett's
* Any history of hypersensitivity to risperidone, or its excipients in formulation, or other known drug allergy
* Patients who received risperidone within 3 months before screening (except p.r.n. use)
* Patients who did not demonstrate sufficient clinical response to an adequate trial of risperidone treatment in the past (an adequate trial is defined as a period of at least 4 weeks at an adequate dose)
* Neurologic disorder (e.g., Neuroleptic Malignant Syndrome, seizure disorders that are unstable, seizure activity within the past 6 months)
* History of alcohol or substance dependence within 3 months of screening
* Female subject who is pregnant (positive beta-HCG) or breast feeding
* Patients with existing moderate or severe EPS or history of tardive dyskinesia
* Patients who have received an experimental drug or used an experimental medical device within 3 months before the planned start of treatment.

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 96 (Actual)
Dates: Start 2007-12; Primary Completion 2009-09 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.
Locations (20):
- United States (20):
  - Dothan, Alabama
  - Phoenix, Arizona
  - Sacramento, California
  - Santa Ana, California
  - Boca Raton, Florida
  - Miami, Florida
  - Smyrna, Georgia
  - Hoffman Estates, Illinois
  - Naperville, Illinois
  - Lake Charles, Louisiana
  - Manhasset, New York
  - New York, New York
  - Staten Island, New York
  - The Bronx, New York
  - Columbus, Ohio
  - Oklahoma City, Oklahoma
  - Philadelphia, Pennsylvania
  - Houston, Texas
  - Fairfax, Virginia
  - Portsmouth, Virginia

REFERENCES:
- [Derived] Iffland M, Livingstone N, Jorgensen M, Hazell P, Gillies D. Pharmacological intervention for irritability, aggression, and self-injury in autism spectrum disorder (ASD). Cochrane Database Syst Rev. 2023 Oct 9;10(10):CD011769. doi: 10.1002/14651858.CD011769.pub2. PMID 37811711
- [Derived] Kent JM, Hough D, Singh J, Karcher K, Pandina G. An open-label extension study of the safety and efficacy of risperidone in children and adolescents with autistic disorder. J Child Adolesc Psychopharmacol. 2013 Dec;23(10):676-86. doi: 10.1089/cap.2012.0058. PMID 24350813
- [Derived] Kent JM, Kushner S, Ning X, Karcher K, Ness S, Aman M, Singh J, Hough D. Risperidone dosing in children and adolescents with autistic disorder: a double-blind, placebo-controlled study. J Autism Dev Disord. 2013 Aug;43(8):1773-83. doi: 10.1007/s10803-012-1723-5. PMID 23212807
- See also: A Study of the Effectiveness and Safety of Two Doses of Risperidone in the Treatment of Children and Adolescents With Autistic Disorder — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=78&filename=CR014740_CSR.pdf

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Double-blind Period. Oral solution for 6 weeks.
- Risperidone Low Dose: Double-blind Period. Risperidone oral solution 0.125 mg (if <45 kg) or 0.175 mg (if >=45 kg) for 6 weeks.
- Risperidone High Dose: Double-blind Period. Risperidone oral solution 1.25 mg (if <45 kg) or 1.75 mg (if >=45 kg) for 6 weeks.
- Placebo/RIS: Open-label Period. Subjects in the double-blind placebo group who continued into open-label risperidone period. Risperidone oral solution 0.125 mg (if <45 kg) or 0.175 mg (if >=45 kg) for 3 days, 0.25 mg tablet on Day 4, flexible dose in 0.25 mg or 0.5 mg increments every 2 weeks, as clinically indicated, to a maximum dose of 1.25 mg (if <45 kg) or 1.75 mg (if >=45 kg).
- Ris Low Dose/RIS: Open-label Period. Subjects in the double-blind risperidone low dose group who continued into open-label risperidone period. Risperidone oral solution 0.125 mg (if <45 kg) or 0.175 mg (if >=45 kg) for 3 days, 0.25 mg tablet on Day 4, flexible dose in 0.25 mg or 0.5 mg increments every 2 weeks, as clinically indicated, to a maximum dose of 1.25 mg (if <45 kg) or 1.75 mg (if >=45 kg).
- Ris High Dose/RIS: Open-label Period. Subjects in the double-blind risperidone high dose group who continued into open-label risperidone period. Risperidone oral solution 0.125 mg (if <45 kg) or 0.175 mg (if >=45 kg) for 3 days, 0.25 mg tablet on Day 4, flexible dose in 0.25 mg or 0.5 mg increments every 2 weeks, as clinically indicated, to a maximum dose of 1.25 mg (if <45 kg) or 1.75 mg (if >=45 kg).
Period: DOUBLE BLIND
Arm/Group | Placebo | Risperidone Low Dose | Risperidone High Dose | Placebo/RIS | Ris Low Dose/RIS | Ris High Dose/RIS
Started | 35 | 30 | 31 | 0 | 0 | 0
Completed | 27 | 25 | 25 | 0 | 0 | 0
Not Completed | 8 | 5 | 6 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 3 | 0 | 0 | 0
Not completed — OTHER | 0 | 2 | 1 | 0 | 0 | 0
Not completed — Lack of Efficacy | 6 | 1 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 0 | 0 | 0
Period: OPEN LABEL
Arm/Group | Placebo | Risperidone Low Dose | Risperidone High Dose | Placebo/RIS | Ris Low Dose/RIS | Ris High Dose/RIS
Started | 0 | 0 | 0 | 30 (26 of 27 double-blind placebo completers and 4 of 8 placebo non-completers entered open-label.) | 24 (24 of 25 double-blind RIS low dose completers and 0 RIS low dose non-completers entered open-label.) | 25 (All 25 double-blind RIS high dose completers and 0 RIS high dose non-completers entered open-label.)
Completed | 0 | 0 | 0 | 19 | 20 | 17
Not Completed | 0 | 0 | 0 | 11 | 4 | 8
Not completed — Adverse Event | 0 | 0 | 0 | 4 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 2 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0 | 1
Not completed — OTHER | 0 | 0 | 0 | 0 | 0 | 2
Not completed — Lack of Efficacy | 0 | 0 | 0 | 2 | 2 | 3
Not completed — Protocol Violation | 0 | 0 | 0 | 2 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Risperidone Low Dose | Risperidone High Dose | Total
Number analyzed (Participants) | 35 | 30 | 31 | 96
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 35 | 30 | 31 | 96
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.6 (2.57) | 10.2 (3.42) | 9.3 (3.11) | 9.3 (3.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 3 | 12
  Male | 31 | 25 | 28 | 84
Region of Enrollment [Number; unit: participants]
  United States of America | 35 | 30 | 31 | 96
Age Categorical [Number; unit: participants]
  <12 years | 30 | 20 | 24 | 74
  >=12 years | 5 | 10 | 7 | 22

OUTCOME MEASURES:

1. Primary Outcome: Change in Aberrant Behavior Checklist Irritability (ABC-I) Subscale
Description: Measure of irritability symptoms of autism. Score range 0 to 45 (lower score = lesser severity).
Time Frame: Baseline and 6 weeks
Population: All randomized subjects with at least one dose of study medication and both baseline and at least one postbaseline value. For subjects who discontinued, Week 6 data is imputed using the subject's last nonmissing, postbaseline value in the double-blind period (Last Observation Carried Forward [LOCF]).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Risperidone Low Dose | Risperidone High Dose
Number analyzed (Participants) | 34 | 29 | 29
units on a scale | -3.5 (10.67) | -7.4 (8.12) | -12.4 (6.52)
Statistical Analysis 1: Comparison: Placebo vs Risperidone High Dose; A step-down testing procedure was employed with the risperidone high dose versus placebo comparison tested first. If this comparison was significant the risperidone low dose versus placebo comparison would be performed. A clinically relevant difference in the change from baseline on the ABC Irritability subscale was assumed to be 6 with a standard deviation of 8. To achieve 80% power with Type I error rate of 5%, 93 subjects were required; Test type: Superiority or Other; p < 0.001, ANCOVA — Type I error is preserved by the step down procedure, no multiple comparison adjustment is needed. A priori threshold for statistical significance was 0.05; ANCOVA model included factors for treatment group, center (after pooling of small centers), baseline weight stratification, and baseline ABC-I value; Mean Difference (Final Values) = -7.9, 95% CI 2-sided [-12.19 to -3.52], Standard Error of Mean 2.18 — Mean difference is change in Risperidone high dose arm minus change in placebo arm
Statistical Analysis 2: Comparison: Placebo vs Risperidone Low Dose; Test type: Superiority or Other; p = 0.164, ANCOVA — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -3.0, 95% CI 2-sided [-7.36 to 1.27], Standard Error of Mean 2.17 — Mean difference is change in Risperidone low dose arm minus change in placebo arm

2. Secondary Outcome: Number of Participants Who Had at Least 25% Improvement in ABC-I
Description: ABC-I is a measure of irritability symptoms of autism with score range 0 to 45 (lower score = lesser severity).
Time Frame: 6 weeks
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Placebo | Risperidone Low Dose | Risperidone High Dose
Number analyzed (Participants) | 34 | 29 | 29
participants | 14 | 15 | 24
Statistical Analysis 1: Comparison: Placebo vs Risperidone High Dose; Test type: Superiority or Other; p = 0.004, Cochran-Mantel-Haenszel — P-value is not adjusted for multiple comparisons; Cochran-Mantel-Haenszel test controlling for center (after pooling small centers) and baseline weight stratification
Statistical Analysis 2: Comparison: Placebo vs Risperidone Low Dose; Test type: Superiority or Other; p = 0.817, Cochran-Mantel-Haenszel — P-value is not adjusted for multiple comparisons; Cochran-Mantel-Haenszel test controlling for center (after pooling small centers) and baseline weight stratification

3. Secondary Outcome: Change in Clinical Global Impression Severity (CGI-S)
Description: Investigator evaluation of severity of illness and functional impairment on a 7-point scale (1="not ill", 2="very mild", 3="mild", 4="moderate", 5="marked", 6="severe", 7="extremely severe").
Time Frame: Baseline and 6 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Risperidone Low Dose | Risperidone High Dose
Number analyzed (Participants) | 34 | 29 | 29
units on a scale | -0.3 (0.79) | -0.4 (0.73) | -1.0 (0.78)
Statistical Analysis 1: Comparison: Placebo vs Risperidone High Dose; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is not adjusted for multiple comparisons; ANCOVA model included factors for treatment group, center (after pooling of small centers), baseline weight stratification, and baseline CGI-S value; Mean Difference (Final Values) = -0.7, 95% CI 2-sided [-1.02 to -0.33], Standard Error of Mean 0.17 — Mean difference is change in Risperidone high dose arm minus change in placebo arm
Statistical Analysis 2: Comparison: Placebo vs Risperidone Low Dose; Test type: Superiority or Other; p = 0.769, ANCOVA — P-value is not adjusted for multiple comparisons; [statistical method as in outcome 3, analysis 1]; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-0.39 to 0.29], Standard Error of Mean 0.17 — Mean difference is change in Risperidone low dose arm minus change in placebo arm

4. Secondary Outcome: Number of Participants Who Had Clinical Global Impression Change Ratings of Much or Very Much Improved.
Description: Investigator impression of change over time from double-blind baseline on a 7-point scale (1="very much improved", 2="much improved", 3="minimally improved", 4="no change", 5="minimally worse", 6="much worse", 7="very much worse").
Time Frame: 6 weeks
Population: All randomized subjects with at least one dose of study medication and at least one postbaseline value. For subjects who discontinued, Week 6 data is imputed using the subject's last nonmissing, postbaseline value in the double-blind period (Last Observation Carried Forward [LOCF]).
Measure: Number; unit: participants
Arm/Group | Placebo | Risperidone Low Dose | Risperidone High Dose
Number analyzed (Participants) | 34 | 30 | 30
participants | 5 | 5 | 19
Statistical Analysis 1: Comparison: Placebo vs Risperidone High Dose; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — P-value is not adjusted for multiple comparisons; Cochran-Mantel-Haenszel test controlling for center (after pooling small centers) and baseline weight stratification
Statistical Analysis 2: Comparison: Placebo vs Risperidone Low Dose; Test type: Superiority or Other; p = 0.985, Cochran-Mantel-Haenszel — P-value is not adjusted for multiple comparisons; Cochran-Mantel-Haenszel test controlling for center (after pooling small centers) and baseline weight stratification

5. Secondary Outcome: Change in Fasting Glucose (mg/dL) at 6 Weeks
Time Frame: Baseline and 6 weeks
Population: All randomized subjects with at least one dose of study medication and both baseline and at least one postbaseline fasting laboratory samples. For subjects who discontinued, Week 6 data is imputed using the subject's last nonmissing, postbaseline value in the double-blind period (Last Observation Carried Forward [LOCF]).
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | Risperidone Low Dose | Risperidone High Dose
Number analyzed (Participants) | 22 | 23 | 23
mg/dL | -0.4 (8.20) | -0.1 (8.81) | -0.3 (9.74)

6. Secondary Outcome: Change in Insulin Resistance (IR) at 6 Weeks
Description: Insulin resistance calculated using the homeostatic model assessment 1 (HOMA1)formula: fasting glucose (mmol/L) times fasting insulin (uU/L) divided by 22.5. HOMA-IR is a widely used clinical tool for estimating insulin resistance based upon the balance between glucose output and insulin secretion. Normal values should be close to 1, while an increase indicates a decrease in insulin sensitivity (or increase in insulin resistance), a potential predictor for the development of Type 2 Diabetes Mellitus.
Time Frame: Baseline and 6 weeks
Population: All randomized subjects with >=1 dose of study medication and fasting glucose and insulin at baseline and at >=1 postbaseline time point. For subjects who discontinued, Week 6 data is imputed using the subject's last nonmissing, postbaseline value in the double-blind period. Means are adjusted for baseline weight (<45 kg, >=45 kg) and baseline IR.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | Risperidone Low Dose | Risperidone High Dose
Number analyzed (Participants) | 22 | 21 | 22
units on a scale | 0.36 [-0.34 to 1.07] | -0.10 [-0.76 to 0.55] | 0.45 [-0.18 to 1.08]

7. Secondary Outcome: Change in Fasting Glucose (mg/dL) at 6 Months
Time Frame: Baseline and 6 months
Population: All subjects with at least one dose of study medication in the open label phase and both double-blind baseline and at least one open-label period fasting laboratory samples. For subjects who discontinued, Month 6 data is imputed using the subject's last nonmissing, postbaseline value in the open-label period.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo/RIS | Ris Low Dose/RIS | Ris High Dose/RIS
Number analyzed (Participants) | 19 | 16 | 16
mg/dL | 4.0 (12.27) | 3.5 (12.26) | 2.3 (8.70)

8. Secondary Outcome: Change in Insulin Resistance (IR) at 6 Months
Description: Insulin resistance calculated using the homeostatic model assessment 1 (HOMA1) formula: fasting glucose (mmol/L) times fasting insulin (uU/L) divided by 22.5. HOMA-IR is a widely used clinical tool for estimating insulin resistance based upon the balance between glucose output and insulin secretion. Normal values should be close to 1, while an increase indicates a decrease in insulin sensitivity (or increase in insulin resistance), a potential predictor for the development of Type 2 Diabetes Mellitus.
Time Frame: Baseline and 6 months
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo/RIS | Ris Low Dose/RIS | Ris High Dose/RIS
Number analyzed (Participants) | 19 | 16 | 16
units on a scale | 0.09 (2.67) | 0.36 (0.89) | 0.75 (0.91)

ADVERSE EVENTS:
Time Frame: Double-blind period: 6 weeks. Open-label period: 6 months.
Groups:
- Open-label Risperidone: Subjects who continued into open-label risperidone period. Risperidone oral solution 0.125 mg (if <45 kg) or 0.175 mg (if >=45 kg) for 3 days, 0.25 mg tablet on Day 4, flexible dose in 0.25 mg or 0.5 mg increments every 2 weeks, as clinically indicated, to a maximum dose of 1.25 mg (if <45 kg) or 1.75 mg (if >=45 kg).
Arm/Group | Placebo | Risperidone Low Dose | Risperidone High Dose | Open-label Risperidone
Serious Adverse Events (participants affected / at risk) | 1/35 | 0/30 | 0/31 | 1/79
Other Adverse Events (participants affected / at risk) | 20/35 | 12/30 | 27/31 | 39/79
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=35) | Risperidone Low Dose (N=30) | Risperidone High Dose (N=31) | Open-label Risperidone (N=79)
Aggression (Psychiatric disorders) | 1 | 0 | 0 | 0
Hydrocele (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=35) | Risperidone Low Dose (N=30) | Risperidone High Dose (N=31) | Open-label Risperidone (N=79)
Abdominal discomfort (Gastrointestinal disorders) | 3 | 0 | 0 | 2
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 2 | 1
Aggression (Psychiatric disorders) | 2 | 0 | 0 | 2
Agitation (Psychiatric disorders) | 2 | 0 | 1 | 3
Akathisia (Nervous system disorders) | 1 | 0 | 2 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 2 | 3
Depression (Psychiatric disorders) | 0 | 0 | 2 | 0
Ear infection (Infections and infestations) | 0 | 0 | 2 | 1
Enuresis (Renal and urinary disorders) | 0 | 2 | 2 | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0
Headache (Nervous system disorders) | 4 | 2 | 2 | 4
Hypersomnia (Nervous system disorders) | 1 | 0 | 2 | 0
Increased appetite (Metabolism and nutrition disorders) | 2 | 5 | 11 | 9
Insomnia (Psychiatric disorders) | 2 | 0 | 0 | 3
Nasopharyngitis (Infections and infestations) | 2 | 2 | 4 | 5
Nausea (Gastrointestinal disorders) | 1 | 1 | 2 | 0
Psychomotor hyperactivity (Nervous system disorders) | 2 | 1 | 1 | 1
Pyrexia (General disorders) | 0 | 0 | 2 | 6
Rash (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 3
Sedation (Nervous system disorders) | 0 | 1 | 8 | 6
Somnolence (Nervous system disorders) | 1 | 0 | 7 | 4
Thirst (General disorders) | 0 | 0 | 2 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 1 | 3 | 6
Vomiting (Gastrointestinal disorders) | 2 | 2 | 2 | 7
Weight increased (Investigations) | 2 | 3 | 4 | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 4
Diarrhea (Gastrointestinal disorders) | 1 | 1 | 0 | 4
Fatigue (General disorders) | 0 | 0 | 1 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can embargo results from a PI's center until the combined results from the completed study have been published in full or the sponsor confirms there will be no multicenter study publication. Results communications must be provided to the sponsor for review at least 60 days before submission for publication. By written request, the sponsor can extend the embargo up to an additional 60 days. The sponsor cannot require changes to scientific content and cannot further extend the embargo.